CLINICAL TRIAL: NCT00000997
Title: Pharmacokinetics and Bioavailability of Dideoxycytidine in Patients With Human Immunodeficiency Virus Infection
Brief Title: A Study of Dideoxycytidine in HIV-Infected Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: ACTG 011; 10987 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Zalcitabine; Drug Evaluation; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Biological Availability
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Zalcitabine

INTERVENTIONS:
Drug: Zalcitabine

SUMMARY:
To determine how much of a dose is absorbed by the body when zalcitabine ( dideoxycytidine; ddC ) is given orally and how long the drug stays in the body after absorption or intravenous (IV) administration.

Laboratory tests have shown that ddC is effective in stopping the growth of the HIV in test tubes. The study will reveal the pharmacokinetic (blood levels) properties of this new drug and how long the drug remains in the body at each of six doses. This should be useful background information and should allow a simple and efficient comparative study of any new oral formulation, such as a tablet or capsule, since dose-related problems will already be known.

DETAILED DESCRIPTION:
Laboratory tests have shown that ddC is effective in stopping the growth of the HIV in test tubes. The study will reveal the pharmacokinetic (blood levels) properties of this new drug and how long the drug remains in the body at each of six doses. This should be useful background information and should allow a simple and efficient comparative study of any new oral formulation, such as a tablet or capsule, since dose-related problems will already be known.

Patients are hospitalized and receive ddC twice, once by mouth and once by IV injection. Each patient receives the drug at one of six increasing doses, and no patient is studied at more than one dose level. Following each dose, toxicity is measured before the next higher dose is given. Several blood samples and urine specimens are taken to permit measurement of the amount of drug in the bloodstream and of the speed with which it is eliminated from the body.

ELIGIBILITY:
Inclusion Criteria

Prior Medication:

Allowed:

* Oral nonabsorbable antifungal agents.

Exclusion Criteria

* Active drug or alcohol abuse.

Co-existing Condition:

* Patients with fever > 102 degrees F at study entry will be excluded.
* Patients with fever > 102 degrees F at study entry will be excluded.

Prior Medication: Excluded:

* Chronic systemic medications.
* Any other experimental drug within 2 weeks of study entry.
* Drugs with known nephrotoxic or hepatotoxic effects within 2 weeks of study entry.
* Drugs known to cause neutropenia within 2 weeks of study entry.
* Rifampin or rifampin derivatives, phenytoin, or barbiturates within 2 weeks of study entry.
* Any other medication except oral nonabsorbable antifungal agents within 72 hours of study entry.

All medications, including aspirin, must be approved by investigator. All medications, including aspirin, must be approved by investigator.

Patients must demonstrate the following clinical and laboratory findings:

* AIDS, AIDS related complex (ARC), or persistent generalized lymphadenopathy as defined by the CDC classification.
* No ascites.
* Off all medications except oral antifungal, nonabsorbable agents for 72 hours prior to study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12
Dates: Study Completion 1988-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lietman P, Study Chair
Locations (1):
- Johns Hopkins Hosp, Baltimore, Maryland, United States

REFERENCES:
- [Background] Gustavson LE, Fukuda EK, Rubio FA, Dunton AW. A pilot study of the bioavailability and pharmacokinetics of 2',3'-dideoxycytidine in patients with AIDS or AIDS-related complex. J Acquir Immune Defic Syndr (1988). 1990;3(1):28-31. PMID 2152803